CLINICAL TRIAL: NCT06236048
Title: Energetics and Glutamate in Schizophrenia
Acronym: EAGLES
Status: Recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 328488
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples for metabolic, mitochondrial markers, glutamate pathways and to determine antipsychotic plasma levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy volunteers
  Interventions: Procedure: MRI scan; Procedure: PET-MR scan
- Schizophrenia - remission
  Interventions: Procedure: MRI scan; Procedure: PET-MR scan
- Treatment resistant schizophrenia
  Interventions: Procedure: MRI scan; Procedure: PET-MR scan

INTERVENTIONS:
Procedure: MRI scan — 7 Tesla MRI scan
Procedure: PET-MR scan — 18F-fluorodeoxyglucose PET-MR scan

SUMMARY:
The goal of this case-control study is to compare brain glutamate, glucose utilisation, lactate production and brain activity in healthy volunteers and people with a diagnosis of schizophrenia.

It investigates the following main questions:

Whether, compared to healthy volunteers, participants with schizophrenia show:

1. reduction in brain glucose utilisation
2. increased brain lactate
3. greater variability in brain glutamate

Participants will be asked to have a screening visit, a MRI brain scan and a PET-MRI brain scan.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteer group:

1. No history of psychiatric illness, as assessed on the Mini neuropsychiatric Interview (MINI).

Treatment responsive schizophrenia group:

1. Meeting ICD-11 criteria for schizophrenia (F20)
2. Meeting symptomatic consensus criteria for remission, defined as scores of mild or less on items P1, P2, P3, N1, N4, N6, G5 and G9 of the PANSS and no history of symptomatic relapse in the past 6 months.
3. Currently receiving one or more of the following antipsychotic medications: Olanzapine; Risperidone; Quetiapine; Amisulpride; Aripiprazole; Paliperidone.
4. Antipsychotic adherent, defined as having a score of >=moderate adherence on the Kemp scale.

Treatment-resistant schizophrenia group:

1. Meeting ICD-11 criteria for schizophrenia (F20)
2. Meeting modified consensus criteria for treatment resistance, including history of at least two antipsychotic treatment trials each lasting ≥6 weeks at a dose of ≥400mg chlorpromazine equivalents.
3. Total PANSS total score > 70
4. Moderate functional impairment (<60 on the SOFAS)
5. Currently receiving one or more of the following antipsychotic medications: Clozapine; Olanzapine; Risperidone; Quetiapine; Amisulpride; Aripiprazole; Paliperidone.
6. Antipsychotic adherent, defined as having a score of >=moderate adherence on the Kemp scale.

Exclusion Criteria:

All participants:

1. Pregnancy or breastfeeding
2. Lacking in mental capacity to provide informed consent to study participation.

2. Diabetes or history of taking an antidiabetic medication 3. Presence of contraindication to MRI at 7 Tesla, including metallic or electronic implants and dental wires.

4. Severe claustrophobia prohibiting participation on PET or MRI 5. Body size above the comfortable limits for the MRI scanner. 6. Previous participation in research or clinical procedure/s involving ionising radiation, which, including the current study, would result in total radiation exposure >=10mSv within 12 months 7. History of head injury resulting in loss of consciousness for > 5 minutes 8. Meeting ICD-11 criteria for organic mental disorder (F00-F09) 9. Meeting ICD-11 criteria for mental and behavioural disorders due to psychoactive substance use (F10-F19) 10. With exclusion of nicotine or cannabis, meeting ICD-11 criteria for psychoactive substance dependence 11. Participation in clinical trial investigating any pharmacological agent other than a licensed antipsychotic compound in the last month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers - community sample people with a diagnosis of schizophrenia - clinical mental health teams.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Brain glucose utilisation | 1 day
  Measured using fully quantitative 18F-fluorodeoxyglucose PET (CMRglc)
Glutamate - anterior cingulate cortex | 1 day
  Glutamate and glutamine measured using magnetic resonance spectroscopy at 7 Tesla
Lactate - visual cortex | 1 day
  Measured using magnetic resonance spectroscopy at 7 Tesla at rest and during visual stimulation
Cerebral blood flow | 1 day
  Measured using arterial spin labelling, 3 Tesla MRI
Cortical network activity | 1 day
  Network activity / connectivity as measured using fMRI at 3 Tesla

CONTACTS AND LOCATIONS:
Locations (1):
- South London and the Maudsley NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
After the end of the study pseudoanonymised data will be available to other researchers.
Supporting Information: Study Protocol
Time Frame: After the primary analyses are completed and published.